CLINICAL TRIAL: NCT01444781
Title: Evaluation of Antibody Persistence Following a Primary Series at 2, 4, and 6 Months on Trial A3L24 and Booster Effect of the DTaP-IPV-Hep B-PRP~T Combined Vaccine or Infanrix Hexa™ Concomitantly Administered With Prevenar™ at 12 to 24 Months of Age in Healthy Latin American Infants
Brief Title: Study of the Booster Effect of DTaP-IPV-Hep B-PRP~T Combined Vaccine or Infanrix Hexa™ and Prevenar™ in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A3L27; U1111-1112-8473 (Other: WHO)
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis
Keywords: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Pediatric combined vaccine; Invasive Hib infections
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis | interventions — Heptavalent Pneumococcal Conjugate Vaccine; HibTITER protein, Haemophilus influenzae; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study Group 1 (Experimental): Participants previously primed with DTaP-IPV-Hep B-PRP~T, will receive one dose of DTaP-IPV-Hep B-PRP~T vaccine + one dose of Prevenar™
  Interventions: Biological: DTaP-IPV-Hep B-PRP~T combined vaccine + Pneumococcal polysaccharide
- Study Group 2 (Active Comparator): Participants previously primed with DTaP-IPV-Hep B-PRP~T, will receive one dose of Infanrix hexa™ vaccine + one dose of Prevenar™
  Interventions: Biological: DTaP-Hep B-IPV // Hib Vaccine + Pneumococcal polysaccharide
- Study Group 3 (Experimental): Participants previously primed with Infanrix hexa™ will receive one dose of DTaP-IPV-Hep B-PRP~T + one dose of Prevenar™.
  Interventions: Biological: DTaP-IPV-Hep B-PRP~T + Pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: DTaP-IPV-Hep B-PRP~T combined vaccine + Pneumococcal polysaccharide — 0.5 mL, Intramuscular each into the right and left deltoid muscle
  Other Names: DTaP-IPV-Hep B-PRP~T vaccine; Prevenar™
  Arms: Study Group 1
Biological: DTaP-Hep B-IPV // Hib Vaccine + Pneumococcal polysaccharide — 0.5 mL, Intramuscular each into the right and left deltoid muscle
  Other Names: Infanrix hexa™; Prevenar™
  Arms: Study Group 2
Biological: DTaP-IPV-Hep B-PRP~T + Pneumococcal polysaccharide vaccine — 0.5 mL (each), Intramuscular each into the right and left deltoid muscle
  Other Names: DTaP-IPV-Hep B-PRP~T combined vaccine; Prevenar™
  Arms: Study Group 3

SUMMARY:
This is a follow-up of the primary series vaccination schedule in Study A3L24 (NCT01177722). The objectives are:

* To describe the antibody persistence to any antigen contained in the investigational DTaP-IPV-Hep B-PRP-T vaccine and Infanrix hexa™ prior to the booster dose
* To describe the safety and immunogenicity of the booster dose of either DTaP-IPV-Hep B-PRP-T or Infanrix hexa™ vaccine.
* To describe the immunogenicity of a booster dose of Prevenar™ given at 12 to 24 months.

DETAILED DESCRIPTION:
All participants who completed trial A3L24 (NCT01177722) will be recruited to participate in this trial. Those who received DTaP-IPV-Hep B-PRP-T combined vaccine will be randomized to receive either a booster dose of DTaP-IPV-Hep B-PRP-T or Infanrix hexa™ vaccine.

Those who received Infanrix hexa™ will receive a booster dose of DTaP-IPV-Hep B-PRP-T combined vaccine. All participants will receive a booster dose of Prevenar™ concomitantly.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 24 months on the day of inclusion.
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative (and by an independent witness(es) if required by local regulations).
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures.
* Toddlers previously included in Study A3L24 who completed the three-dose primary series vaccination of either DTaP-IPV-Hep B-PRP~T or Infanrix hexa™ at 2,4 and 6 months of age according to protocol (both concomitantly administered with Prevenar™ and Rotarix™).

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the booster vaccinations.
* Planned participation in another clinical trial during the present trial period.
* Receipt of any vaccine in the 4 weeks preceding the booster vaccinations, except in case of pandemic influenza vaccination, which may be received at least two weeks before the study vaccines.
* Planned receipt of any vaccine in the 4 weeks following the trial vaccinations.
* Previous booster vaccination against pertussis, tetanus, diphtheria, poliomyelitis, Haemophilus influenzae type b, hepatitis B and pneumococcal infection(s) with either the trial vaccine or another vaccine.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 3 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Laboratory-confirmed or clinical suspicion of personal or maternal seropositivity for Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C, as reported by the parent/guardian.
* History of pertussis, tetanus, diphtheria, poliomyelitis, Haemophilus influenzae type b, hepatitis B and pneumococcal infection(s), confirmed either clinically, serologically, or microbiologically.
* At high risk for opportunistic infection during the trial.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances.
* History of contraindication to receipt of pertussis-containing vaccine.
* Laboratory-confirmed or clinical suspicion of thrombocytopenia contraindicating Intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* History of seizures .
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Receipt of oral or injected antibiotic therapy within 72 hours prior to the first blood draw
* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1106 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- Cali, Colombia
- San José, Costa Rica

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 26 September 2011 through 19 July 2012 at 2 clinic centers in Colombia and Costa Rica.
Pre-assignment Details: A total of 1106 participants who met all of the inclusion and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of DTaP-IPV-Hep B-PRP~T vaccine and one dose of Prevenar (PCV7)
- Group2: DTaPIPV-Hep B-PRP~T Primary/Infanrix Hexa+PCV7 Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of Infanrix Hexa vaccine and one dose of PCV7.
- Group3: Infanrix Hexa Primary/DTaPIPV-Hep B PRP~T+PCV7 Booster: Participants who were previously primed with Infanrix Hexa vaccine received one dose of DTaP-IPV-Hep B-PRP~T and one dose of PCV7
Period: Overall Study
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group2: DTaPIPV-Hep B-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group3: Infanrix Hexa Primary/DTaPIPV-Hep B PRP~T+PCV7 Booster
Started | 416 | 415 | 275
Completed | 413 | 411 | 272
Not Completed | 3 | 4 | 3
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- DTaP IPV Hep B PRP T + Prevenar™ Primary and Booster Group: Participants who were previously primed with DTaP IPV Hep B PRP T received one dose of DTaP IPV Hep B PRP T vaccine and one dose of Prevenar (PCV7)
- DTaP IPV Hep B PRP T Primary/Infanrix Hexa+PCV7 Booster Group: Participants who were previously primed with DTaP IPV Hep B PRP T received one dose of Infanrix Hexa vaccine and one dose of PCV7.
- Infanrix Hexa Primary/DTaP IPV Hep B PRP T+PCV7 Booster Group.: Participants who were previously primed with Infanrix Hexa vaccine received one dose of DTaP IPV Hep B PRP T and one dose of PCV7
- Total: Total of all reporting groups
Arm/Group | DTaP IPV Hep B PRP T + Prevenar™ Primary and Booster Group | DTaP IPV Hep B PRP T Primary/Infanrix Hexa+PCV7 Booster Group | Infanrix Hexa Primary/DTaP IPV Hep B PRP T+PCV7 Booster Group. | Total
Number analyzed (Participants) | 416 | 415 | 275 | 1106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 416 | 415 | 275 | 1106
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.6 (3.25) | 17.6 (3.34) | 17.8 (3.26) | 17.7 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 186 | 128 | 517
  Male | 213 | 229 | 147 | 589
Region of Enrollment [Number; unit: Participants]
  Colombia | 266 | 266 | 172 | 704
  Costa Rica | 150 | 149 | 103 | 402

OUTCOME MEASURES:

1. Primary Outcome: Summary of Diphtheria and Tetanus Post Primary Series Antibodies, Persistence and Booster Response Following Vaccination With Either DTaP-IPV Hep B-PRP T Vaccine or Infanrix Hexa Vaccine
Description: Anti-Diphtheria (D) antibodies were measured by a toxin neutralization test. Anti-Tetanus (T) antibodies were measured by enzyme-linked immunosorbent assay (ELISA). Antibody persistence for anti-Diphtheria and anti-Tetanus antibodies was defined as titers ≥0.01 IU/mL and ≥0.1 IU/mL before the booster dose at Day 0. Booster response to Diphtheria and Tetanus was defined as antibody titers ≥0.01 IU/mL and ≥0.1 IU/mL at Day 30 post-booster vaccination.
  Day 140 = Primary series; Day 0 = Pre-booster; and Day 30 = Post-booster titers
Time Frame: Day 140 (Primary series) and Day 0 (Pre-booster)
Population: Antibody responses were assessed in the Per Protocol Analysis Set, which includes all persons who did not have any protocol deviations.
Measure: Number; unit: Participants
Groups:
- Group 1: DTaP IPV Hep B PRP T + Prevenar™ Primary and Booster: Participants who were previously primed with DTaP IPV Hep B PRP T received one dose of DTaP IPV Hep B PRP T vaccine and one dose of Prevenar (PCV7)
- Group 2DTaP IPV Hep B PRP T Primary/Infanrix Hexa+PCV7 Booster: Participants who were previously primed with DTaP IPV Hep B PRP T received one dose of Infanrix Hexa vaccine and one dose of PCV7.
- Group 3Infanrix Hexa Primary/DTaP IPV Hep B PRP T+PCV7 Booster: Participants who were previously primed with Infanrix Hexa vaccine received one dose of DTaP IPV Hep B PRP T and one dose of PCV7
Arm/Group | Group 1: DTaP IPV Hep B PRP T + Prevenar™ Primary and Booster | Group 2DTaP IPV Hep B PRP T Primary/Infanrix Hexa+PCV7 Booster | Group 3Infanrix Hexa Primary/DTaP IPV Hep B PRP T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Participants
  Anti-Diphtheria Day140 ≥0.01 IU/mL (N=392,391,259) | 392 | 391 [0 to 0] | 259 [0 to 0]
  Anti-Diphtheria Day 140 ≥0.1 IU/mL (N=392,391,259) | 308 | 290 [0 to 0] | 197 [0 to 0]
  Anti-Diphtheria Day 0 ≥0.01 IU/mL (N=390,390,257) | 382 | 378 [0 to 0] | 246 [0 to 0]
  Anti-Diphtheria Day 0 ≥0.1 IU/mL (N=390,390,257) | 156 | 153 [0 to 0] | 70 [0 to 0]
  Anti-Diphtheria Day 30 ≥0.01 IU/mL (N=393,387,254) | 393 | 387 [0 to 0] | 254 [0 to 0]
  Anti-Diphtheria Day 30 ≥0.1 IU/mL (N=393,387,254) | 393 | 386 [0 to 0] | 254 [0 to 0]
  Anti-Tetanus Day 140 ≥0.01 IU/mL (N=392,391,258) | 392 | 391 [0 to 0] | 258 [0 to 0]
  Anti-Tetanus Day 140 ≥0.1 IU/mL (N=392,391,258) | 392 | 390 [0 to 0] | 258 [0 to 0]
  Anti-Tetanus Day 0 ≥0.01 IU/mL (N=389,387,255) | 389 | 386 [0 to 0] | 255 [0 to 0]
  Anti-Tetanus Day 0 ≥0.1 IU/mL (N=389,387,255) | 289 | 286 [0 to 0] | 196 [0 to 0]
  Anti-Tetanus Day 30 ≥0.01 IU/mL (N=392,385,254) | 392 | 385 [0 to 0] | 254 [0 to 0]
  Anti-Tetanus Day 30 ≥0.1 IU/mL (N=392,385,254) | 391 | 385 [0 to 0] | 254 [0 to 0]

2. Primary Outcome: Summary of Pertussis and Filamentous Haemagglutinin Post Primary Series Antibodies, Persistence and Booster Response Following Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine
Description: Anti-Pertussis toxin (PT) and anti-Filamentous haemagglutinin (FHA) antibodies were measured by ELISA. Antibody persistence for anti-PT and anti-FHA was defined as titers ≥ lower limit of quantitation (LLOQ) before the booster dose at Day 0. Booster responses for PT and FHA at Day 30 were defined as: pre-vaccination antibody concentrations < LLOQ and post-vaccination levels ≥ 4 x LLOQ, pre-vaccination antibody concentrations ≥ LLOQ but < 4 x LLOQ and post/pre vaccination ≥ 4, and pre-vaccination antibody concentrations ≥ 4 x LLOQ and post/pre-vaccination ≥ 2.
  Day 140 = Primary series; Day 0 = Pre-booster; and Day 30 = Post-booster titers.
Time Frame: Day 140 after primary vaccination, Day 0 (pre-vaccination), and Day 30 after final booster vaccination
Population: Antibody responses were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Groups:
- Group 1: DTaP-IPV Hep B-PRP~T + Prevenar™ Primary and Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of DTaP-IPV-Hep B-PRP~T vaccine and one dose of Prevenar (PCV7)
- Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of Infanrix Hexa vaccine and one dose of PCV7.
- Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster: Participants who were previously primed with Infanrix Hexa vaccine received one dose of DTaP-IPV-Hep B-PRP~T and one dose of PCV7
Arm/Group | Group 1: DTaP-IPV Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Participants
  Anti-PT Day 140 ≥2 EU/mL (N=393,391,259) | 393 | 391 [0 to 0] | 259 [0 to 0]
  Anti-PT Day 0 ≥2 EU/mL (N=385,382,257) | 344 | 349 [0 to 0] | 225 [0 to 0]
  A-PT Day 30 ≥ 2 EU/mL (N=391,383,254) | 391 | 383 [0 to 0] | 254 [0 to 0]
  Anti-PT 4-fold increase (N=380,374,252) | 353 | 351 [0 to 0] | 234 [0 to 0]
  Anti-PT booster response (N=380,374,252) | 375 | 365 [0 to 0] | 245 [0 to 0]
  Anti-FHA Day 140 ≥2 EU/mL (N=391,390,259) | 391 | 390 [0 to 0] | 259 [0 to 0]
  Anti-FHA Day 0 ≥2 EU/mL (N=389,384,255) | 389 | 384 [0 to 0] | 253 [0 to 0]
  Anti-FHA Day 30 ≥2 EU/mL (N=390,385,254) | 390 | 385 [0 to 0] | 254 [0 to 0]
  Anti-FHA 4-fold increase (N=384,376,252) | 336 | 334 [0 to 0] | 235 [0 to 0]
  Anti-FHA booster response (N=384,376,252) | 370 | 367 [0 to 0] | 249 [0 to 0]

3. Primary Outcome: Summary of Polio Antibodies Post Primary Series, Persistence and Booster Response Following Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine
Description: Anti-Poliovirus types 1, 2, and 3 antibodies were measured by neutralization assay. Antibody persistence for anti-Poliovirus 1, 2, and 3 was defined as antibody titers ≥8 (1/dil) before the booster dose at Day 0. Booster response to Poliovirus 1, 2, and 3 was defined as antibody titers ≥8 (1/dil) at Day 30.
  Day 140 = Primary series; Day 0 = Pre-booster; and Day 30 = Post-booster titers.
Time Frame: Day 140 after primary vaccination, Day 0 (pre-vaccination), and Day 30 after final booster vaccination
Population: Antibody responses were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP IPV Hep B PRP T + Prevenar™ Primary and Booster | Group 2DTaP IPV Hep B PRP T Primary/Infanrix Hexa+PCV7 Booster | Group 3Infanrix Hexa Primary/DTaP IPV Hep B PRP T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Participants
  Anti-Polio 1 Day 140 (N = 338,329,214) | 338 | 329 [0 to 0] | 214 [0 to 0]
  Anti-Polio 1 Day 0 (N = 338,326,213) | 334 | 320 [0 to 0] | 210 [0 to 0]
  Anti-Polio 1 Day 30 (N = 339,327,212) | 339 | 327 [0 to 0] | 212 [0 to 0]
  Anti-Polio 2 Day 140 (N = 338,327,214) | 338 | 327 [0 to 0] | 214 [0 to 0]
  Anti-Polio 2 Day 0(N = 337,328,213) | 335 | 328 [0 to 0] | 213 [0 to 0]
  Anti-Polio 2 Day 30 (N = 340,327,212) | 340 | 327 [0 to 0] | 212 [0 to 0]
  Anti-Polio 3 Day 140 (N = 338,328,214) | 338 | 328 [0 to 0] | 214 [0 to 0]
  Anti-Polio 3 Day 0 (N = 338,326,213) | 324 | 309 [0 to 0] | 211 [0 to 0]
  Anti-Polio 3 Day 30 (N = 340,326,212) | 340 | 326 [0 to 0] | 212 [0 to 0]

4. Primary Outcome: Summary of Hepatitis B and Haemophilus Influenzae Type B Post Primary Series Antibodies; Antibody Persistence, and Booster Response Following Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine
Description: Anti-Hepatitis B antibodies were measured by the commercially available VITROS ECi/ECiQ Immunodiagnostic System. Anti-Haemophilus influenza type b capsular polyribosyl ribitol phosphate (PRP) antibodies were measured using a Farr type radioimmunoassay that used radiolabeled PRP (3H PRP) in the presence of 36Cl (volume marker). Anti-Hepatitis antibody titers ≥ 10 mIU/mL and ≥ 100 mIU/mL at Day 0 confirmed antibody persistence and booster response at Day 30. Anti-PRP antibody titers ≥ 0.15 µg/ml and ≥ 1.0 µg/ml at Day 0 confirmed antibody persistence and booster response at Day 30.
  Day 140 = Primary series; Day 0 = Pre-booster; and Day 30 = Post-booster titers.
Time Frame: Day 140 after primary vaccination, Day 0 (pre-vaccination), and Day 30 after final booster vaccination
Population: Antibody responses were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Participants
  Anti-Hep B Day 140 ≥10 mIU/mL (N = 393,392,260) | 391 | 391 [0 to 0] | 260 [0 to 0]
  Anti-Hep B Day 140 ≥100 mIU/mL (N = 393,392,260) | 389 | 387 [0 to 0] | 259 [0 to 0]
  Anti-Hep B Day 0 ≥10 mIU/mL (N = 396,391,259) | 386 | 382 [0 to 0] | 257 [0 to 0]
  Anti-Hep B Day 0 ≥100 mIU/mL (N = 396,391,259) | 327 | 333 [0 to 0] | 213 [0 to 0]
  Anti-Hep B Day 30 ≥10 mIU/mL (N = 395,393,259) | 394 | 391 [0 to 0] | 259 [0 to 0]
  Anti-Hep B Day 30 ≥100 mIU/mL (N = 395,393,259) | 386 | 384 [0 to 0] | 257 [0 to 0]
  Anti-PRP Day 140 ≥0.15 µg/mL (N = 393,392,260) | 370 | 375 [0 to 0] | 246 [0 to 0]
  Anti-PRP Day 140 ≥1.0 µg/mL (N = 393,392,260) | 297 | 305 [0 to 0] | 188 [0 to 0]
  Anti-PRP Day 0 ≥0.15 µg/mL (N = 395,391,258) | 290 | 304 [0 to 0] | 197 [0 to 0]
  Anti-PRP Day 0 ≥1.0 µg/mL (N = 395,391,258) | 110 | 129 [0 to 0] | 73 [0 to 0]
  Anti-PRP Day 30 ≥0.15 µg/mL (N = 396,391,258) | 395 | 391 [0 to 0] | 258 [0 to 0]
  Anti-PRP Day 30 ≥1.0 µg/mL (N = 396,391,258) | 391 | 387 [0 to 0] | 258 [0 to 0]

5. Secondary Outcome: Summary of Geometric Mean Titers to Vaccine Antibodies Post Primary Vaccination Series; Before and After Booster Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine.
Description: Anti-Diphtheria antibodies were measured by a toxin neutralization test. Anti-Tetanus, anti-PT, and anti-FHA antibodies were measured by ELISA. Anti-Poliovirus types 1, 2, and 3 were measured by neutralization assay. Anti-Hepatitis B antibodies were measured by the commercially available VITROS ECi/ECiQ Immunodiagnostic System. Anti-PRP antibodies were measured using a Farr type radioimmunoassay that used radiolabeled PRP (3H PRP) in the presence of 36Cl (volume marker).
  Day 140 = Primary series; Day 0 = Pre-booster; and Day 30 = Post-booster titers.
Time Frame: Day 140 after primary vaccination, Day 0 (pre-vaccination), and Day 30 after final booster vaccination
Population: Geometric mean titers against vaccine antibodies were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP IPV Hep B PRP T + Prevenar™ Primary and Booster | Group 2DTaP IPV Hep B PRP T Primary/Infanrix Hexa+PCV7 Booster | Group 3Infanrix Hexa Primary/DTaP IPV Hep B PRP T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Titers
  Anti-Diphtheria Day 140 (N=392,391,259) | 0.265 [0.237 to 0.295] | 0.254 [0.227 to 0.285] | 0.251 [0.220 to 0.286]
  Anti-Diphtheria Day 0 (N=390,390,257) | 0.077 [0.069 to 0.086] | 0.074 [0.066 to 0.083] | 0.059 [0.051 to 0.068]
  Anti-Diphtheria Day 30 (N=393,387,254) | 5.55 [5.07 to 6.08] | 4.40 [3.99 to 4.86] | 6.05 [5.41 to 6.76]
  Anti-Tetanus Day 140 (N=392,391,258) | 1.50 [1.39 to 1.61] | 1.54 [1.44 to 1.65] | 1.80 [1.68 to 1.93]
  Anti-Tetanus Day 0 (N=389,387,255) | 0.208 [0.188 to 0.231] | 0.224 [0.200 to 0.251] | 0.201 [0.180 to 0.225]
  Anti-Tetanus Day 30 (N=392,385,254) | 5.72 [5.21 to 6.27] | 5.21 [4.78 to 5.68] | 7.52 [6.63 to 8.52]
  Anti-PT Day 140 (N=393,391,259) | 99.6 [94.0 to 106] | 102 [96.6 to 108] | 97.0 [90.1 to 105]
  Anti-PT Day 0 (N=385,382,257) | 7.43 [6.63 to 8.32] | 8.47 [7.52 to 9.56] | 7.41 [6.38 to 8.61]
  Anti PT D30 (N=391,383,254) | 154 [143 to 166] | 191 [178 to 206] | 140 [127 to 153]
  Anti-FHA Day 140 (N=391,390,259) | 179 [169 to 190] | 187 [176 to 199] | 120 [112 to 129]
  Anti-FHA Day 0 (N=389,384,255) | 21.2 [18.9 to 23.8] | 23.4 [20.8 to 26.3] | 14.4 [12.5 to 16.8]
  Anti-FHA Day 30 (N=390,385,254) | 316 [293 to 342] | 418 [386 to 454] | 260 [231 to 293]
  Anti-Polio 1 Day 140 (N=338,329,214) | 656 [587 to 734] | 705 [625 to 796] | 1276 [1098 to 1484]
  Anti-Polio 1 Day 0 (N=338,326,213) | 132 [116 to 150] | 134 [116 to 154] | 224 [188 to 267]
  Anti-Polio 1 Day 30 (N=339,327,212) | 2140 [1937 to 2364] | 2633 [2363 to 2933] | 2978 [2592 to 3421]
  Anti-Polio 2 Day 140 (N=338,327,214) | 1152 [1035 to 1282] | 1241 [1101 to 1398] | 1945 [1676 to 2256]
  Anti-Polio 2 Day 0 (N=337,328,213) | 251 [214 to 294] | 289 [245 to 341] | 380 [313 to 461]
  Anti-Polio 2 Day 30 (N=340,327,212) | 4232 [3821 to 4688] | 4887 [4372 to 5463] | 6369 [5569 to 7283]
  Anti-Polio 3 Day 140 (N=338,328,214) | 1169 [1025 to 1332] | 1108 [979 to 1255] | 1948 [1647 to 2304]
  Anti-Polio 3 Day 0 (N=338,326,213) | 128 [109 to 149] | 126 [106 to 150] | 207 [173 to 248]
  Anti-Polio 3 Day 30 (N=340,326,212) | 3569 [3164 to 4027] | 3322 [2939 to 3755] | 6015 [5244 to 6898]
  Anti-Hepatitis B Day 140 (N=393,392,260) | 3050 [2715 to 3427] | 3180 [2834 to 3568] | 2910 [2556 to 3313]
  Anti-Hepatitis B Day 0 (N=396,391,259) | 386 [332 to 449] | 406 [349 to 472] | 336 [284 to 397]
  Anti-Hepatitis B Day 30 (N=395,393,259) | 8462 [7154 to 10010] | 11218 [9482 to 13272] | 9688 [7940 to 11821]
  Anti-PRP Day 140 (N=393,392,260) | 3.19 [2.69 to 3.78] | 3.60 [3.05 to 4.25] | 2.13 [1.78 to 2.54]
  Ant-PRP Day 0 (N=395,391,258) | 0.482 [0.406 to 0.573] | 0.556 [0.472 to 0.656] | 0.455 [0.375 to 0.553]
  Anti-PRP Day 30 (N=396,391,258) | 42.4 [37.0 to 48.6] | 41.5 [36.6 to 47.0] | 56.5 [48.4 to 65.9]

6. Secondary Outcome: Summary of Immune Response Against Serotypes in the Prevenar Vaccine After Booster Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine
Description: Anti-Streptococcus pneumococcal type specific antibody (anti-Pn PS) was measured by ELISA. Booster response to pneumococcal serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F was defined as antibody titers ≥0.35 µg/mL at Day 30.
Time Frame: Day 30 after final booster vaccination
Population: Antibody responses against Prevenar vaccine serotypes were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Groups:
- Group 2:DTaP-IPV-HepB PRP~T Primary/Infanrix Hexa+PCV7 Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of Infanrix Hexa vaccine and one dose of PCV7.
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Participants
  Anti-Pneumococcal 4 (N=161,147,94) | 160 | 146 [0 to 0] | 94 [0 to 0]
  Anti-Pneumococcal 6B (N=160,146,94) | 155 | 145 [0 to 0] | 93 [0 to 0]
  Anti-Pneumococcal 9V (N=161,147,94) | 161 | 147 [0 to 0] | 94 [0 to 0]
  Anti-Pneumococcal 14 (N=161,147,94) | 161 | 147 [0 to 0] | 94 [0 to 0]
  Anti-Pneumococcal 18C (N=161,147,94) | 160 | 147 [0 to 0] | 94 [0 to 0]
  Anti-Pneumococcal 19F (N=161,147,94) | 161 | 144 [0 to 0] | 94 [0 to 0]
  Anti-Pneumococcal 23F (N=158,145,93) | 158 | 144 [0 to 0] | 93 [0 to 0]

7. Secondary Outcome: Summary of Geometric Mean Titers to Prevenar Vaccine Antibodies After Booster Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine
Description: Anti-Streptococcus pneumococcal type specific antibody (anti-Pn PS) was measured by ELISA.
Time Frame: Day 30 after final booster vaccination
Population: Geometric mean titers against Prevenar vaccine serotypes were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Titers
  Anti-Pneumococcal 4 (N=161,147,94) | 2.79 [2.47 to 3.15] | 3.03 [2.64 to 3.47] | 3.58 [3.07 to 4.17]
  Anti-Pneumococcal 6B (N=160,146,94) | 6.87 [5.68 to 8.31] | 8.98 [7.86 to 10.3] | 9.34 [7.76 to 11.2]
  Anti-Pneumococcal 9V (N=161,147,94) | 2.51 [2.22 to 2.85] | 2.86 [2.57 to 3.19] | 2.92 [2.50 to 3.42]
  Anti-Pneumococcal 14 (N=161,147,94) | 11.6 [10.2 to 13.2] | 13.2 [11.5 to 15.2] | 12.3 [10.2 to 14.7]
  Anti-Pneumococcal 18C (N=161,147,94) | 2.37 [2.10 to 2.67] | 2.63 [2.35 to 2.95] | 3.40 [2.92 to 3.94]
  Anti-Pneumococcal 19F (N=161,147,94) | 3.01 [2.62 to 3.47] | 3.74 [3.19 to 4.38] | 3.72 [3.19 to 4.32]
  Anti-Pneumococcal 23F (N=158,145,93) | 6.98 [6.14 to 7.94] | 7.20 [6.23 to 8.33] | 9.30 [7.79 to 11.1]

8. Secondary Outcome: Summary of Booster Response to Vaccine Antigens Before and After Booster Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine By Age Strata
Description: Anti-PT and anti-FHA antibodies were measured by ELISA.
Time Frame: Day 0 (pre-vaccination) and Day 30 after final booster vaccination
Population: Booster responses to vaccine antigens were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Participants
  Anti-PT ≥12 to <15 month Day 0 (N=104,105,61) | 100 | 104 [0 to 0] | 61 [0 to 0]
  Anti-PT ≥12 to <15 moth Day 30 4-fold N=103,102,60 | 87 | 92 [0 to 0] | 53 [0 to 0]
  Anti-PT ≥12 to <15 months Booster (N=103,102,60) | 100 | 99 [0 to 0] | 56 [0 to 0]
  Anti-PT ≥15 to <19 month Day 0 (N=142,128,96) | 133 | 118 [0 to 0] | 86 [0 to 0]
  Anti-PT ≥15 to <19 moth Day 30 4-fold N=140,126,95 | 132 | 121 [0 to 0] | 89 [0 to 0]
  Anti-PT ≥15 to <19 month Booster (N=140,126,95) | 138 | 125 [0 to 0] | 94 [0 to 0]
  Anti-PT ≥19 to ≤24 months Day 0 (N=139,149,100) | 111 | 127 [0 to 0] | 78 [0 to 0]
  AntiPT ≥19 to ≤24 month Day 30 4 fold N=137,146,97 | 134 | 138 [0 to 0] | 92 [0 to 0]
  Anti-PT ≥19 to ≤24 months Booster (N=137,146,97) | 136 | 141 [0 to 0] | 95 [0 to 0]
  Anti-FHA ≥12 to <15 months Day 0 (N=103,105,59) | 103 | 105 [0 to 0] | 59 [0 to 0]
  Anti-FHA ≥12 to <15 mos Day 30 4-fold N=103,101,58 | 76 | 78 [0 to 0] | 53 [0 to 0]
  Anti-FHA ≥12 to <15 months Booster (N=103,101,58) | 96 | 99 [0 to 0] | 58 [0 to 0]
  Anti-FHA ≥15 to <19 month Day 0 (N=143,130,96) | 143 | 130 [0 to 0] | 95 [0 to 0]
  Anti-FHA ≥15 to <19 mos Day 30 4-fold N=140,128,96 | 127 | 118 [0 to 0] | 88 [0 to 0]
  Anti-FHA ≥15 to <19 months Booster (N=140,128,96) | 136 | 124 [0 to 0] | 94 [0 to 0]
  Anti-FHA ≥19 to ≤24 month Day 0 (N=143,149,100) | 143 | 149 [0 to 0] | 99 [0 to 0]
  Anti-FHA ≥19 to ≤24 mos Day 30 4-fold N=141,147,98 | 133 | 138 [0 to 0] | 94 [0 to 0]
  Anti-FHA ≥19 to ≤ 24 months Booster (N=141,147,98) | 138 | 144 [0 to 0] | 97 [0 to 0]

9. Secondary Outcome: Summary of Geometric Mean Titers to Vaccine Antigens After Booster Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine by Age Strata
Description: Anti-Diphtheria antibodies were measured by a toxin neutralization test. Anti-FHA antibodies were measured by ELISA. Anti-Poliovirus types 1, 2, and 3 were measured by neutralization assay.
Time Frame: Day 30 after final booster vaccination
Population: Geometric mean titers to vaccine antigens were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 396 | 393 | 260
Titers
  Anti-Diphtheria ≥12 to <15 months (N=103,107,59) | 3.20 [2.72 to 3.76] | 2.73 [2.30 to 3.24] | 3.82 [3.01 to 4.84]
  Anti-Diphtheria ≥15 to <19 months (N=144,129,95) | 6.39 [5.56 to 7.34] | 4.77 [3.98 to 5.72] | 6.56 [5.43 to 7.92]
  Anti-Diphtheria ≥19 to ≤24 months (N=146,151,100) | 7.14 [6.17 to 8.26] | 5.77 [5.00 to 6.66] | 7.34 [6.30 to 8.56]
  Anti-FHA ≥12 to <15 months (N=103,105,60) | 235 [209 to 263] | 268 [233 to 308] | 197 [156 to 248]
  Anti-FHA ≥15 to <19 months (N=143,130,96) | 339 [294 to 392] | 453 [392 to 524] | 280 [236 to 331]
  Anti-FHA ≥19 to ≤24 months (N=144,150,98) | 365 [322 to 414] | 533 [473 to 599] | 287 [232 to 356]
  Anti-Polio 3 ≥12 to <15 months (N=87,92,45) | 2509 [1944 to 3240] | 2616 [2098 to 3263] | 5617 [4006 to 7876]
  Anti-Polio 3 ≥15 to <19 months (N=128,114,81) | 3944 [3265 to 4764] | 3261 [2585 to 4113] | 5409 [4359 to 6713]
  Anti-Polio 3 ≥19 to ≤24 months (N=125,120,86) | 4119 [3398 to 4993] | 4061 [3387 to 4869] | 6889 [5583 to 8499]

10. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions Following Booster Vaccination With Either DTaP-IPV-Hep B-PRP~T Vaccine or Infanrix Hexa Vaccine
Description: Solicited injection site: Pain, Erythema, Swelling, and Extensive swelling of vaccinated limb; Solicited systemic reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability. Grade 3 Injection site: Pain, Cries if limb is moved or reduced movement; Erythema and Swelling, ≥5 cm; Extensive swelling of limb, Severe. Grade 3 Systemic reactions: Pyrexia (Temperature) >39.5˚C; Vomiting, ≥ 6 times per 24 hours or needing parenteral nutrition; Crying, >3 hours; Somnolence, Sleeping often or difficulty waking; Anorexia, refuses ≥3 meals; and Irritability, Inconsolable.
Time Frame: Day 0 up to Day 7 after final booster vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set, which includes all persons who received the study or control vaccine.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 416 | 415 | 275
Participants
  Injection site Pain (N=413,412,272) | 232 | 205 [0 to 0] | 160 [0 to 0]
  Grade 3 inj. site Pain (N=413,412,272) | 10 | 6 | 6
  Injection site Erythema (N=413,412,272) | 112 | 100 [0 to 0] | 86 [0 to 0]
  Grade 3 inj. site Erythema (N=413,412,272) | 4 | 3 | 7
  Injection site Swelling (N=412,412,272) | 60 | 56 [0 to 0] | 49 [0 to 0]
  Grade 3 inj. site Swelling (N=412,412,272) | 3 | 3 | 1
  Extensive swelling of limb (N=413,412,272) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Extensive swelling of limb (N=413,412,272) | 0 | 0 | 0
  Pyrexia (N=413,412,272) | 114 | 99 [0 to 0] | 91 [0 to 0]
  Grade 3 Pyrexia (N=413,412,272) | 2 | 6 | 1
  Vomiting (N=413,412,272) | 34 | 39 [0 to 0] | 19 [0 to 0]
  Grade 3 Vomiting (N=413,412,272) | 1 | 1 | 0
  Crying (N=413,412,272) | 148 | 139 [0 to 0] | 102 [0 to 0]
  Grade 3 Crying (N=413,412,272) | 1 | 1 | 2
  Somnolence (N=413,412,272) | 124 | 113 [0 to 0] | 85 [0 to 0]
  Grade 3 Somnolence (N=413,412,272) | 2 | 1 | 2
  Anorexia (N=413,412,272) | 118 | 121 [0 to 0] | 90 [0 to 0]
  Grade 3 Anorexia (N=413,412,272) | 3 | 3 | 4
  Irritability (N=413,412,272) | 201 | 176 [0 to 0] | 146 [0 to 0]
  Grade 3 Irritability (N=413,412,272) | 1 | 3 | 2

11. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site Following Booster Vaccination With Prevenar Vaccine
Description: Solicited injection site: Pain, Erythema, Swelling, and Extensive swelling of vaccinated limb. Grade 3 Injection site: Pain, cries if limb is moved or reduced movement; Erythema and Swelling, ≥5 cm; and Extensive swelling of limb, Severe.
Time Frame: Day 0 up to Day 7 after final booster vaccination
Population: Solicited injection site reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Groups:
- Group 1: DTaP-IPV-Hep B-PRP~ T + Prevenar™ Primary and Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of DTaP-IPV-Hep B-PRP~T vaccine and one dose of Prevenar (PCV7)
- Group 2: DTaP-IPV-HepB-PRP~Tprimary/Infanrix Hexa+PCV7 Booster: Participants who were previously primed with DTaP-IPV-Hep B-PRP~T received one dose of Infanrix Hexa vaccine and one dose of PCV7.
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~ T + Prevenar™ Primary and Booster | Group 2: DTaP-IPV-HepB-PRP~Tprimary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Number analyzed (Participants) | 416 | 415 | 275
Participants
  Injection site Pain (N=413,412,272) | 224 | 184 [0 to 0] | 140 [0 to 0]
  Grade 3 Injection site Pain (N=413,412,272) | 9 | 9 | 5
  Injection site Erythema (N=413,412,272) | 84 | 77 [0 to 0] | 52 [0 to 0]
  Grade 3 Injection site Erythema (N=413,412,272) | 0 | 0 | 0
  Injection site Swelling (N=413,412,272) | 51 | 42 [0 to 0] | 33 [0 to 0]
  Grade 3 Injection site Swelling (N=413,412,272) | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 30 after final booster vaccination.
Description: The total number (N) for solicited adverse events in the table reflects those participants for which the diary cards were returned and for which data were available for the event during the period.
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster
Serious Adverse Events (participants affected / at risk) | 13/416 | 15/415 | 9/275
Other Adverse Events (participants affected / at risk) | 253/416 | 221/415 | 168/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster (N=416) | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster (N=415) | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster (N=275)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Kawasaki's disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: DTaP-IPV-Hep B-PRP~T + Prevenar™ Primary and Booster (N=416) | Group 2:DTaP-IPV-HepB-PRP~T Primary/Infanrix Hexa+PCV7 Booster (N=415) | Group 3:Infanrix Hexa Primary/DTaP-IPV-HepB-PRP~T+PCV7 Booster (N=275)
Nasopharyngitis (Infections and infestations) | 27 (27) | 23 (23) | 12 (12)
Injection site Pain (General disorders) | 232 (232) | 205/412 (205) | 160/272 (160)
Injection site Erythema (General disorders) | 112/413 (112) | 100/412 (100) | 86/272 (86)
Injection site Swelling (General disorders) | 60/412 (60) | 56/412 (56) | 49/272 (49)
Pyrexia (General disorders) | 114/413 (114) | 99/412 (99) | 91/272 (91)
Vomiting (Gastrointestinal disorders) | 34/413 (34) | 39/412 (39) | 19/272 (19)
Crying (Psychiatric disorders) | 148/413 (148) | 139/412 (139) | 102/272 (102)
Drowsiness (Nervous system disorders) | 124/413 (124) | 113/412 (113) | 85/272 (85)
Anorexia (Metabolism and nutrition disorders) | 118/413 (118) | 121/412 (121) | 90/272 (90)
Irritability (Psychiatric disorders) | 201/413 (201) | 176/412 (176) | 146/272 (146)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.